CLINICAL TRIAL: NCT03622749
Title: Pilot Study of Neuromodulation for Enhancement of Emotion Regulation in Bipolar Mood Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Kristen K. Ellard, Ph.D., Instructor in Psychology, Massachusetts General Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2018P001227; 1T32NS100663-01 (NIH)
Record Dates: First submitted 2018-07-11; First posted 2018-08-09 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2024-02

CONDITIONS: Bipolar Disorder; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Bipolar Disorder | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Patients (Active Comparator): Individuals with Bipolar 1 Disorder
  Interventions: Device: Transcranial Magnetic Stimulation (TMS)
- Controls (No Intervention): Healthy controls

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation (TMS) — Non-Invasive neuromodulation
  Arms: Patients

SUMMARY:
The investigators are conducting this research study to better understand how individuals with bipolar disorder regulate their emotions, and if the study can use a technique called "transcranial magnetic stimulation" or TMS to help improve emotion regulation for individuals with bipolar disorder.

DETAILED DESCRIPTION:
Emotion dysregulation contributes to the development and maintenance of a wide range of psychopathology, but is especially relevant for individuals with bipolar mood disorders (BD). These individuals experience severe and episodic emotion dysregulation associated with maladaptive functioning, interpersonal problems, decreased work productivity, and suicidal ideation and behavior. To date, both pharmacological and psychosocial treatments fail to normalize emotion dysregulation for many bipolar patients. As a consequence, all too many experience poor outcomes. Thus, there is a significant need for new innovative approaches to target and improve emotion dysregulation in bipolar patients. Non-invasive neuromodulation using transcranial magnetic stimulation (TMS) may provide a viable strategy to help improve emotion dysregulation in bipolar mood disorders. As a first step to test this hypothesis, the current proposal seeks to experimentally identify specific neural target sites for improving emotion regulation using TMS. If the investigators can demonstrate target engagement of emotion regulation at the behavioral level using TMS, this will provide an important first step towards examining the potential utility of TMS as a viable strategy to help improve emotion dysregulation in bipolar mood disorders. While this is not a definitive clinical trial, the sham-controlled double-crossover design of this study will provide valuable information for target site selection for the development of TMS as an intervention strategy to improve emotion dysregulation in BD.

ELIGIBILITY:
Inclusion Criteria:

* Patients

  * Men and women
  * Ages 18-50 years
  * Patients diagnosed with bipolar I disorder (BD-I), current mood state euthymic.
  * On a stable psychiatric medication regimen for at least a month prior to and during study participation

Healthy Controls:

* Men and women
* Ages 18-50 years
* Without major psychiatric illness

Exclusion Criteria:

* Patients

  * Any change in psychiatric medications within a month prior to and during study participation
  * Legal or mental incompetency
  * Intellectual disability
  * Current manic (YMRS > 12) or severe depressive episode (HAM-D-17 > 5)
  * Substance use disorder (abuse or dependence) with active use within the last 3 months
  * Significant medical or neurological illness
  * Prior neurosurgical procedure
  * History of seizures
  * History of ECT treatment or clinical TMS within the past three months
  * Implanted cardiac pacemakers
  * Patients who have conductive, ferromagnetic or other magnetic-sensitive metals implanted in their head or neck, or are non-removable and within 30 cm of the treatment coil. These include:

    * Aneurysm clips or coils
    * Carotid or cerebral stents
    * Metallic devices implanted in the head (e.g. Implanted pacemaker, medication pump, vagal stimulator, deep brain stimulator, TENS unit, or ventriculo-peritoneal shunt)
    * Magnetically active dental implants
    * Cochlear/otologic implants
    * CSF shunts
    * Ferromagnetic ocular implants
    * Pellets, bullets, fragments less than 30 cm from the coil
    * Facial tattoos with metallic ink, permanent makeup less than 30 cm from the coil
  * Pregnant women

Healthy Controls:

* History of major psychiatric illness, including psychosis
* Has a first-degree relative with psychosis
* Active use of neuropsychoactive medications
* Legal or mental incompetency
* Intellectual disability
* Substance use disorder (abuse or dependence) with active use within the last 3 months
* Significant medical or neurological illness
* Prior neurosurgical procedure
* History of seizures
* History of ECT treatment or clinical TMS within the past three months
* Implanted cardiac pacemakers
* Individuals who have conductive, ferromagnetic or other magnetic-sensitive metals implanted in their head or neck, or are non-removable and within 30 cm of the treatment coil. These include:

  * Aneurysm clips or coils
  * Carotid or cerebral stents
  * Metallic devices implanted in the head (e.g. Implanted pacemaker, medication pump, vagal stimulator, deep brain stimulator, TENS unit, or ventriculo-peritoneal shunt)
  * Magnetically active dental implants
  * Cochlear/otologic implants
  * CSF shunts
  * Ferromagnetic ocular implants
  * Pellets, bullets, fragments less than 30 cm from the coil
  * Facial tattoos with metallic ink, permanent makeup less than 30 cm from the coil
* Pregnant women

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Change Emotion Conflict Resolution Task | Change from baseline to 15 minutes post-TMS stimulation
  Slope of reaction time (milliseconds)
Change Cognitive Reappraisal Task | Change from baseline to 15 minutes post-TMS stimulation
  Distress rating (scale 1- 4)

CONTACTS AND LOCATIONS:
Overall Officials: Kristen K Ellard, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Martinos Center for Biomedical Imaging, Charlestown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No